CLINICAL TRIAL: NCT03221465
Title: Project LIFT - Lifestyle Intervention to Promote Fitness in Transplantation
Brief Title: Project LIFT - Promoting Healthy Behavior Through a Wearable Fitness Device and Financial Incentives
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 825784
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Kidney Transplant; Complications; Liver Transplant; Complications; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Principal Investigators are neither given names of particular participants nor assignment to study arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Usual care: dietary and exercise counseling only at baseline, no other intervention.
- Usual Care + self-monitoring of physical activity (Active Comparator): Tracking Device control: The intervention applied is usual care and self-monitoring of physical activity. Patients will receive a pedometer (e.g. Misfit brand wrist pedometer) to allow for self-monitoring of physical activity. They will be able to obtain daily feedback on step counts via the wearable device and their smartphones. They will also have a 2-week run-in period like the incentive arm.
  Interventions: Behavioral: Usual care and self-monitoring of physical activity
- Self-monitoring + incentives of physical activity (Experimental): The intervention applied is self-monitoring of physical activity with incentives. Patients will receive a a pedometer (e.g. Misfit brand wrist pedometer) to allow for self-monitoring of physical activity. Participants will monitor daily step counts with automated feedback on goal attainment via text message. We will establish a baseline step count for each participant (during a 2-week run-in period) and then recommend a 15 percentage point increase in daily step goal every 2 weeks during the 12-week intervention period (weeks 3-14) with a maximum goal of 7,000 steps. Two health engagement questions will be sent per week to participants as well for the 12-week intervention period.
  Interventions: Behavioral: Self-monitoring of physical activity with incentives

INTERVENTIONS:
Behavioral: Self-monitoring of physical activity with incentives — Participants are given a pedometer (e.g. Misfit brand wrist pedometer) to allow self-monitoring of physical activity and receive financial incentives. Participants also answer two health questions a week for 12 weeks.
  Arms: Self-monitoring + incentives of physical activity
Behavioral: Usual care and self-monitoring of physical activity — Participants simply given a pedometer (e.g. Misfit brand wrist pedometer) with no other intervention to allow self-monitoring of physical activity.
  Arms: Usual Care + self-monitoring of physical activity

SUMMARY:
Project LIFT is a randomized, controlled trial that tests the effectiveness of a remotely-monitored, home-based exercise program utilizing wearable fitness trackers to monitor steps taken per day, health engagement questions, and financial incentives. 120 subjects will be randomized into 3 arms: 1) usual care - no fitness tracker or incentive, 2) a fitness tracker + no incentives, and 3) fitness tracker plus financial incentives.

DETAILED DESCRIPTION:
Obesity is the most common diseases in the United States - an estimated 35% of adults are obese. Among kidney (KT) and liver transplant (LT) recipients, weight gain and obesity is associated with poor graft function. Yet, within a year of transplantation, habituation to a sedentary lifestyle, changes in metabolism, and immunosuppression drugs contribute to an average 4-10 kg weight gain for recipients. Recent innovations in wearable device technology can passively monitor an individual's physical activity. Additionally, incentives and health questions designed using insights from behavioral economics have been shown to motivate device engagement and improvements in health behaviors. A remotely-monitored exercise program could improve behavior change and potentially be durable because it takes advantage of the high motivation for improving health in this population. The objective of this study is to use a randomized, controlled trial to test the efficacy of a home-based exercise program using wearable devices, health engagement questions and financial incentives. Participants in the intervention arm will establish a baseline step count during the first two weeks, followed by a 12-week intervention period and a 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Kidney transplant, Liver transplant, Simultaneous liver-kidney, or kidney-pancreas transplant recipients at the Hospital of the University of Pennsylvania within 2-24 months of transplantation
2. Ability to read and provide informed consent in English to participate in the study
3. Possess a smartphone with a data plan and willing to receive text messages
4. Willing to walk and sync wearable daily during the 2-week run-in in order to determine baseline [for Arms 2 & 3]
5. Willing to provide a final weight at study end.

Exclusion Criteria:

1. Inability to provide informed consent
2. Does not have daily access to a smartphone compatible with the wearable device
3. Unable or unwilling to complete the baseline measurements and survey, or perform the exit interview and weigh-in
4. Already enrolled in a financial incentive-based exercise program using a wearable device
5. Use of a wearable accelerometer or pedometer outside of the study protocol for step-tracking; (e.g., Fitbit; using phone step-tracker is acceptable; using existing wearable for cycling or swimming is acceptable)
6. Any other medical conditions that would prohibit participation in a physical activity program
7. Severe vision, hearing, or mobility impairment precluding participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Final Weight | End of 4 month study period
  Weight of patient at end of 4 month period of study.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Serper, MD, Principal Investigator — University of Pennsylvania Hospital System
Locations (2):
- United States (2):
  - Northwestern University Comprehensive Transplant Center, Chicago, Illinois
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Galanti G, Stefani L, Mascherini G, Petri C, Corsani I, Francini L, Cattozzo A, Gianassi M, Minetti E, Pacini A, Cala PG. Short-term prospective study of prescribed physical activity in kidney transplant recipients. Intern Emerg Med. 2016 Feb;11(1):61-7. doi: 10.1007/s11739-015-1294-5. Epub 2015 Sep 4. PMID 26341217
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- [Background] Richards J, Gunson B, Johnson J, Neuberger J. Weight gain and obesity after liver transplantation. Transpl Int. 2005 Apr;18(4):461-6. doi: 10.1111/j.1432-2277.2004.00067.x. PMID 15773968
- [Background] Patel MS, Asch DA, Volpp KG. Wearable devices as facilitators, not drivers, of health behavior change. JAMA. 2015 Feb 3;313(5):459-60. doi: 10.1001/jama.2014.14781. No abstract available. PMID 25569175
- [Background] Case MA, Burwick HA, Volpp KG, Patel MS. Accuracy of smartphone applications and wearable devices for tracking physical activity data. JAMA. 2015 Feb 10;313(6):625-6. doi: 10.1001/jama.2014.17841. No abstract available. PMID 25668268
- [Background] Tudor-Locke C, Hatano Y, Pangrazi RP, Kang M. Revisiting "how many steps are enough?". Med Sci Sports Exerc. 2008 Jul;40(7 Suppl):S537-43. doi: 10.1249/MSS.0b013e31817c7133. PMID 18562971